CLINICAL TRIAL: NCT03059667
Title: A Randomized Non-comparative Phase II Study of Anti-PDL1 ATEZOLIZUMAB (MPDL3280A) or Chemotherapy as Second-line Therapy in Patients With Small Cell Lung Cancer (SCLC)
Brief Title: Immunotherapy as Second-line in Patient With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1603
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Small Cell Lung Cancer; Small Cell Lung Cancer Limited Stage; Small Cell Lung Cancer Extensive Stage
Keywords: Small Cell Lun cancer; IFCT; immune therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Topotecan; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : chemotherapy (Active Comparator): Patients randomly assigned to the control arm will receive either:
  * topotecan (oral 2.3 mg/m² or IV 1.5 mg/m² day 1-4 recommended)
  * or re-induction by carboplatin - etoposide chemotherapy.
  Interventions: Drug: Topotecan; Drug: Carboplatin; Drug: Etoposide
- Arm B : immune therapy (Experimental): Patients randomly assigned to the experimental arm will receive Anti PDL1 ATEZOLIZUMAB (MPDL3280A) at a fixed dose of 1200 mg IV every three weeks until progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab at 1200 mg IV every 3 weeks
  Arms: Arm B : immune therapy
Drug: Topotecan — oral 2.3 mg/m² or IV 1.5 mg/m² day 1-4 recommended
  Arms: Arm A : chemotherapy
Drug: Carboplatin — In accordance with the summary of product characteristics.
  Arms: Arm A : chemotherapy
Drug: Etoposide — In accordance with the summary of product characteristics.
  Arms: Arm A : chemotherapy

SUMMARY:
Chemotherapy still constitutes the backbone of small-cell lung cancer (SCLC) therapy, particularly in the extensive disease (ED) stage (ED-SCLC). Despite the fact that a substantial complete response rate could be achieved in SCLC patients receiving etoposide - cisplatin doublet, cure remains the exception. Overall survival in patients receiving this combination is 10 months and progression free survival 6.3 months. At time of progression two options are hitherto accepted: reinduction of carboplatin - etoposide doublet or, for patients unfit for reinduction, topotecan single-drug regimen. However, in both clinical cases, median survival hardly achieves 33 weeks. Consistent data using anti - PDL1 (Programmed death-ligand 1) or anti PD1 (programmed cell death 1) antibodies suggest that they are active as single drug regimens in many malignant diseases. Taking into account the rich tumor infiltrating lymphocyte in pathological specimens of SCLC, we can hypothesize that experimental use of ATEZOLIZUMAB (MPDL3280A) in patients is ethical pending that it demonstrates activity in the second line setting.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed small-cell lung cancer.
2. Extensive or limited disease according to the criteria of the Veteran's Administration Lung Cancer Group: (disease extended is defined as a disease beyond hemi thorax and supraclavicular lymph node areas. Tumor pleural effusion will be considered as extended disease).
3. Targetable tumor lesions according to RECIST 1.1. Tumor involvement encompassed into a radiotherapy field is eligible as target pending that progression is documented.
4. Tumor sample sent to IFCT for PD-L1 immunohistochemistry
5. Previous platinum - etoposide treatment for at least 2 cycles.
6. Demonstrated progression of the disease other than brain metastasis or carcinomatous meningitis.

   For the patient relapsing more than one year after the end of the previous treatment, a new histological confirmation is required before randomization.
7. Age over 18 years.
8. Weight loss ≤ 10% during the last three months.
9. Patients with brain metastases at diagnosis will be eligible pending that they have achieved brain response during the first line therapy (including brain radiotherapy is required) and remain in brain tumor response during the two months prior to randomization.
10. Performance Status 0-2
11. Creatinine clearance > 40 mL/min.
12. Neutrophils ≥ 2,000 µL-1 and platelets ≥ 100,000 µL-1.
13. Bilirubin ≤ 1.5 x normal.
14. Transaminases, alkaline phosphatases ≤ 2.5 x ULN except in case of liver metastases (5 x ULN).
15. Electrocardiogram without sign of progressive coronaropathy.
16. No approved or investigational anti-cancer therapy concurrently or in the 5 years prior to start of study drug except the first line of treatment of the SCLC, including tumor embolization, chemotherapy, radiation therapy, immunotherapy, hormone therapy, biologic therapy, or anti angiogenic therapy (e.g., inhibitors of VEGF or VEGFR (Vascular Endothelial Growth Factor Receptor).
17. Signed informed consent
18. A female is eligible to enter and participate in this study if she is of:

Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has undergone:

* Hysterectomy.
* Bilateral oophorectomy (ovariectomy).
* Bilateral tubal ligation.
* Or who is post-menopausal:
* Patients not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone value >40 mIU/mL and an estradiol value <40 pg/mL (<140 pmol/L).
* Subject using HRT must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH (Follicle Stimulating Hormone) and estradiol concentrations prior to initiation of HRT (Hormone Replacement Therapy).

Childbearing potential, including any female who has had a negative serum pregnancy test within 1 week prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Contraceptive methods acceptable to the IFCT, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

* An intrauterine device with a documented failure rate of less than 1% per year.
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
* Double-barrier contraception: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Oral contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implant of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches The contraceptive methods must be used during all the time of the treatment and must be maintained during 5 months after the end of the treatment in the Atezolizumab arm and 30 days for women, 90 days for men, after the end of the treatment in the chemotherapy arm.

Female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 15 days following the last dose of study drug.

A male with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.

Exclusion Criteria:

1. Non-small cell lung cancer or mixed small-cell lung cancer - non small cell cancer.
2. Prior immunotherapy
3. Last dose of the previous treatment received less than 21 days before randomization (washout period).
4. Corticosteroid with a daily dose over 10 mg prednisolone or equivalent for more than 10 days during the previous month.
5. Unstable angina or uncontrolled cardiac disease.
6. Progressive infection (suggested by a fever associated with hyperleukocytosis, increase procalcitonin, and increase of C reactive protein without link with a paraneoplastic syndrome).
7. Patient not able to follow the therapeutic program.
8. Natremia < 125 mmol/L except in case of corrective treatment before the beginning of the therapy.
9. Hypercalcemia despite corrective treatment (corrected calcemia = Ca++ (mmol) + [(40-alb (g)) x 0.025].
10. Psychic or mental disease that do not allow the patient to give informed consent.
11. Pregnant or lactating female.
12. Systemic immunosuppressive therapy (eg cyclophosphamide, azathioprine, methotrexate, thalidomide and anti-tumor necrosis factor [TNF]) during the two weeks preceding the day 1 of cycle 1.
13. Auto-immune disease. History of autoimmune disease, including myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, syndrome Guillain-Barré, multiple sclerosis, vasculitis or glomerulonephritis. Patients with a history of hypothyroidism origin autoimmune treated with a stable dose replacement therapy may be eligible for this study. Patients with controlled type 1 diabetes treated with insulin are eligible in this study.
14. Idiopathic pulmonary fibrosis history, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced lung disease, idiopathic pulmonary or active signs of pneumonia or interstitial lung infiltrate (any cause) detected on the lung scan selection
15. Prior malignancy. Note: Patients who have had another malignancy and were treated more than 5 years ago and have since been considered cured, or patients with a history of basocellular skin carcinoma or in situ carcinoma of the uterine cervix are eligible.
16. Presence of any concurrent disease or condition that would make the subject inappropriate for study participation including any unresolved or unstable, serious toxicity from prior administration of another investigational drug or any serious medical disorder that would interfere with the subject's safety, obtaining informed consent, or compliance with all study related procedures.
17. Administration of a live attenuated vaccine during the four weeks preceding the day 1 of cycle 1, or administration of a vaccine of this type scheduled during the study. An influenza vaccine should be administered during the influenza season (approximately from October to March). Patients should not receive a live attenuated influenza vaccine during the four weeks preceding the day 1 of cycle 1, and shall not receive a vaccine of this type during the study.
18. History of human immunodeficiency virus infection or chronic hepatitis B or C.
19. Presence of active or uncontrolled infection.
20. Psoriasis patients
21. History of any one or more of the following cardiovascular conditions within the past 6 months:

    * Coronary/peripheral artery bypass graft, cardiac angioplasty or stenting.
    * Myocardial infarction.
    * Severe/unstable angina pectoris.
    * Symptomatic peripheral vascular disease, pulmonary embolism or untreated deep venous thrombosis (DVT), cerebrovascular accident or transient ischemic attack.
    * Note: Subject with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
    * Class III or IV congestive heart failure, as defined by the New York Heart Association.
22. Concurrent treatment with an investigational agent or participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Response Rate in the experimental arm | 6 weeks
  Maximum changed in target lesions from baseline at 6 weeks

SECONDARY OUTCOMES:
Progression Free Survival | approximately 36 weeks
  Progression-free survival is defined as the time from randomization to first observation of progression or date of death (from any cause). Patients who did not progress or not die will be censored on the date of their last tumor assessment, i.e. on the last date that we really know that the patient was considered as "progression free".
Overall Survival | approximately 8 months
  Overall survival, defined as the time from randomization until death due to any cause, will be the principal secondary endpoint. For patients who do not die, time to death will be censored at the time of last contact.
Compliance assessed by the number of cycle received by patient | approximately 36 weeks
Safety assessed by the maximum grade will be summarized by frequency and proportion of total patients, by system organ class and NCI-CTC, Version 4.0 categories. | approximately 36 weeks
  The maximum grade will be summarized by frequency and proportion of total patients, by system organ class and NCI-CTC, Version 4.0 categories.
Duration of response | approximately 36 weeks
Quality of life assessed by scale | approximately 36 weeks

OTHER OUTCOMES:
Response rate according to tissue PD-L1 expression | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PUJOL, MD PhD, Principal Investigator — CHU de Montpellier
Locations (18):
- France (18):
  - Annemasse - CH, Ambilly
  - Angers - CHU, Angers
  - CH, Colmar
  - CHRU Grenoble, Grenoble
  - Centre Hospitalier - Pneumologie, Le Mans
  - Lorient - CHBS, Lorient
  - Montpellier - CHRU, Montpellier
  - Mulhouse - CH, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - APHP - Paris Bichat, Paris
  - GH Paris Saint-Joseph, Paris
  - CHG de Pau, Pau
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Rouen - CHU, Rouen
  - Centre Hospitalier, Saint-Quentin
  - Toulouse - CHU Larrey, Toulouse
  - CHU Tours - Pneumologie, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Negre E, Coffy A, Langlais A, Daures JP, Lavole A, Quoix E, Molinier O, Greillier L, Audigier-Valette C, Moro-Sibilot D, Westeel V, Morin F, Roch B, Pujol JL. Development and Validation of a Simplified Prognostic Score in SCLC. JTO Clin Res Rep. 2020 Feb 12;1(1):100016. doi: 10.1016/j.jtocrr.2020.100016. eCollection 2020 Mar. PMID 34589918
- See also: IFCT website — https://www.ifct.fr/index.php/fr/la-recherche/item/2050-ifct-1603-petites-cellules